CLINICAL TRIAL: NCT01774461
Title: Influence of Remote Ischemic Preconditioning on Cardiac Function After Endurance Exercise
Brief Title: Ischemic Preconditioning in Endurance Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: METC12-2-038
Record Dates: First submitted 2012-07-09; First posted 2013-01-24 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham RIC (No Intervention): Control treatment (sham RIC) will consist of four 5-minute simulated inflations of a blood pressure cuff placed on the upper arm. The inflations will be separated by 5-minute periods when the blood pressure cuff will be deflated.
- Remote ischemic conditioning (Active Comparator): Blood pressure cuff placed on upper arm and inflated to 200mmHg for 5 minutes then deflated for 5 minutes - this cycle is repeated a total of 4 times.
  Interventions: Other: Remote ischemic preconditioning

INTERVENTIONS:
Other: Remote ischemic preconditioning — Blood pressure cuff placed on upper arm and inflated to 200mmHg for 5 minutes then deflated for 5 minutes - this cycle is repeated a total of 4 times.
  Arms: Remote ischemic conditioning

SUMMARY:
The aim of this study is to investigate the effect of remote ischemic preconditioning on biochemical and functional indices of cardiac function induced by a 30 km run in healthy trained long distance runners.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Healthy
* Age between 18 and 65 years
* Endurance-trained (two or more training sessions per week)

Exclusion Criteria:

* Not applicable

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Serum concentrations of cardiac troponins | 6 hours, 2 hourly time intervals

SECONDARY OUTCOMES:
Indices of cardiac function measured by echocardiography | 2 hours post-exercise

CONTACTS AND LOCATIONS:
Overall Officials: Marja van Dieijen-Visser, PhD, Principal Investigator — Department of Clinical Chemistry, MUMC, Maastricht, the Netherlands
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands